CLINICAL TRIAL: NCT04569552
Title: Urdu Version of the Unified PARKINSON Disease Rating Scale: a Reliability and Validity Study
Brief Title: Urdu Version of the Unified PARKINSON Disease Rating Scale
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Collaborators: University of Lahore (Other)
Responsible Party: Sponsor
Other Study IDs: REC-FSD-00227 Muhammad Kashif
Record Dates: First submitted 2020-09-24; First posted 2020-09-30 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; Validity; Reliability; UPDRS
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The Unified Parkinson's Disease Rating Scale version 3.0 (UPDRS), published in 1987, was developed to provide a comprehensive instrument for the evaluation of impairment and disability related to PD. The primary objectives of this research were to translate, validate and generate data on the UPDRS for using among Urdu speaking residents of Pakistan. UPDRS questionnaire will be first translated into Urdu and then apply on Parkinson's Disease patients to check the validity and reliability of this scale . Instrument will be first translated from English to Urdu by two experts. Both these experts were fluent in English and Urdu language.

One expert belongs to allied health care profession and other expert will be junior life scientist. The third expert compares the initial to Urdu translation and formulated the first draft of UPDRS. Content validity of UPDRS Questionnaire was established by committee method. 10 experts from physical therapy field rate the all items of the UPDRS on content validity index . They rate each item of UPDRS Questionnaire for its relevance, clarity, simplicity, and ambiguity on four point ordinal likert scale. Data will be analyzed using SPSS v 25. Intra class correlation coefficient, chronbach alpha and factor analysis will be used to analyses the data.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a complex disorder with a combination of characteristic motor signs and non-motor symptoms. The natural course of PD is modified by the effect of treatments, and over time, these treatments can also be associated with both motor and non-motor complications. At present, there is no biomarker or other gold standard index to determine the severity of PD as a whole. Therefore, measurement of the different aspects of PD and their severities relies on clinically based rating scales.

The Unified Parkinson's Disease Rating Scale version 3.0 (UPDRS), published in 1987, was developed to provide a comprehensive instrument for the evaluation of impairment and disability related to PD. Further, the scale attempted to utilize the most clinically relevant aspects of several earlier scales that were already familiar to clinicians and researchers, though poorly validated clinimetrically. The development of this "unified" scale was aimed to provide a single scale so that outcomes among different clinical trials could be directly compared. For two decades, the UPDRS was the most used scale for assessment of PD patients and became the reference scale for development of other measures and for the United States and European regulatory agencies.

In 2002, the Movement Disorder Society sponsored Task Force for Rating Scales in PD carried out a review and critique of the UPDRS. Several weaknesses, including ambiguities in wording, the absence of uniform instructions for raters, some metric flaws, and the lack of assessments for many important non-motor symptoms were evident. Therefore, a modified UPDRS, named the Movement Disorder Society-UPDRS (MDS-UPDRS), was proposed to overcome the identified shortcomings. In 2008, the official MDS-UPDRS English version was published along with satisfactory clinimetric results on its performance in a series of over 800 native English-speaking patients and raters. As a result, the MDS-UPDRS has been proposed as the official benchmark scale for PD.

Given the content and structure of the MDS-UPDRS, with inclusion of symptoms impossible to assess objectively (e.g., fatigue, pain, dizziness), a questionnaire for self-evaluation, and a wide body of instructions for raters, the scale has to be cross-culturally adapted and validated. A detailed plan for obtaining equivalent and locally validated non-English versions of the MDS-UPDRS was established by the Steering Committee of the Movement Disorder Society Task Force and Spanish, Italian and Estonian official versions are now available.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease.
* Modified Hoehn and Yahr Scale(H&Y stages I to III),
* Independent in transfers
* A score equal to or greater than 24 on the Mini-Mental State Examination (MMSE), and
* Previous lack of participation in balance or motor training.

Exclusion Criteria:

* History of any neurological conditions such as stroke, multiple sclerosis, epilepsy other than Parkinson's disease,
* History of orthopedic issues such as pain, fracture, or lower limb pathology,
* History of visual abnormalities,
* History of any chronic or cardiovascular pathology that can interfere with the transfer procedure or can affect the training sessions,
* The participants having severe dyskinesia or "on-off" phases,
* Previous history of surgery for PD,
* History of virtual games used for treatment in the past three months, and
* Virtual game phobia.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects were at least 50 years of age and were at Hoehn and Yahr stage 3.0 or less. The diagnosis of PD was made by a movement disorders specialist based on the presence of at least two of the three cardinal signs of PD (resting tremor, rigidity, or bradykinesia) without a known or suspected alternative cause of parkinsonism.
Sampling Method: Non-Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
Unified Parkinson's Disease Rating Scale | 1 Week
  UPDRS is a subjective tool with widespread use in the clinical settings used for the Parkinson disease (PD). This scale includes 31 items divided into three sub-scales; sub-scale-I includes scoring on mentation, behavior and mood, sub-scale-II includes scoring on activities of daily living and sub-scale-III assesses motor system. This test predicts the performance of physical performance of the adult population affected with the neurological impairments and the performance comes out to be really well when used in combination with Berg Balance Scale. The test is authenticated to be able to detect minimal changes in performance over time and to be used across variety of rehabilitation interventions. A possible maximum of 199 points can be scored in this scale. 199 score refers to complete disability and 0 refers to absence of disability

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, PhD*, Principal Investigator — University of Lahore
Locations (1):
- University Institute of Physical Therapy, The University of Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siderowf A, McDermott M, Kieburtz K, Blindauer K, Plumb S, Shoulson I; Parkinson Study Group. Test-retest reliability of the unified Parkinson's disease rating scale in patients with early Parkinson's disease: results from a multicenter clinical trial. Mov Disord. 2002 Jul;17(4):758-63. doi: 10.1002/mds.10011. PMID 12210871
- [Background] Movement Disorder Society Task Force on Rating Scales for Parkinson's Disease. The Unified Parkinson's Disease Rating Scale (UPDRS): status and recommendations. Mov Disord. 2003 Jul;18(7):738-50. doi: 10.1002/mds.10473. PMID 12815652
- [Background] Abdolahi A, Scoglio N, Killoran A, Dorsey ER, Biglan KM. Potential reliability and validity of a modified version of the Unified Parkinson's Disease Rating Scale that could be administered remotely. Parkinsonism Relat Disord. 2013 Feb;19(2):218-21. doi: 10.1016/j.parkreldis.2012.10.008. Epub 2012 Oct 25. PMID 23102808
- [Background] Post B, Merkus MP, de Bie RM, de Haan RJ, Speelman JD. Unified Parkinson's disease rating scale motor examination: are ratings of nurses, residents in neurology, and movement disorders specialists interchangeable? Mov Disord. 2005 Dec;20(12):1577-84. doi: 10.1002/mds.20640. PMID 16116612
- [Background] van Hilten JJ, van der Zwan AD, Zwinderman AH, Roos RA. Rating impairment and disability in Parkinson's disease: evaluation of the Unified Parkinson's Disease Rating Scale. Mov Disord. 1994 Jan;9(1):84-8. doi: 10.1002/mds.870090113. PMID 8139609